CLINICAL TRIAL: NCT04545489
Title: A Nurse-led Intervention to Extend the Veteran HIV Treatment Cascade for Cardiovascular Disease Prevention (V-EXTRA-CVD)
Brief Title: A Nurse-led Intervention to Extend the Veteran HIV Treatment Cascade for Cardiovascular Disease Prevention
Acronym: V-EXTRA-CVD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IIR 19-418
Record Dates: First submitted 2020-09-03; First posted 2020-09-11 (Actual); Results first posted 2025-10-30 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Cardiovascular Disease; Hypertension; Care Coordination; HIV Treatment Cascade
Keywords: HIV; Cardiovascular Disease; Medication Management; Care Coordination
MeSH Terms: conditions — Cardiovascular Diseases; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): Participants randomized to the intervention will have 4 visits over 12 months with study staff. In addition, they will also receive focused communication from the interventionist (nurse or pharmacist), with additional BP monitoring support and medication management for 12 months.
  Interventions: Behavioral: Intervention group
- Education control group (Active Comparator): Participants randomized to the education control group will have 4 visits over 12 months and will receive education materials related to CVD risk reduction.
  Interventions: Behavioral: Education control group

INTERVENTIONS:
Behavioral: Intervention group — This is a intervention for 12 months which focuses on behavioral and medication management, led by a health coach (nurse or pharmacist)
  Arms: Intervention group
Behavioral: Education control group — This group will receive education materials related to CVD risk reduction at each 4 month visit over the course of 12 months.
  Arms: Education control group

SUMMARY:
The VA is the largest single provider of HIV care in the US and Veterans with HIV use significantly more healthcare services and have a 1.5-2x higher risk of atherosclerotic cardiovascular disease (ASCVD) compared to uninfected Veterans. The goal is to improve BP treatment for Veterans with HIV to reduce ASCVD risk. Within a randomized controlled trial (RCT), the investigators hypothesize that the VA adapted nurse-led intervention will result in a clinically significant 6 millimeters of mercury (mmHg) reduction in systolic blood pressure (SBP) over 12 months compared to those receiving enhanced education only. The study is innovative because of the use of stakeholder-engaged design process, multi-component nurse-led intervention, and VA Video Connect (VVC) to monitor CVD risk factors. The project meets VA strategic priorities including: 1) greater choice for Veterans; 2) improve timeliness of services; 3) focus more resources more efficiently (strengthen foundational services in VA). If shown to be effective, this intervention will have substantial impact among high-risk Veterans, potentially reducing ASCVD events by more than a quarter.

DETAILED DESCRIPTION:
Background: The VA is the largest provider of HIV care in the United States. The ~31,000 Veterans with HIV use significantly more healthcare and have up to 2x higher risk of atherosclerotic cardiovascular disease (ASCVD) compared to uninfected Veterans. The HIV treatment cascade model includes care steps; once people obtain remission, providers should focus on preventing ASCVD. The investigators will extend the HIV treatment cascade and focus on reducing ASCVD risk among people with HIV. Veterans with HIV have low perceived risk for ASCVD and uptake of guideline-based treatment for BP is low.

Significance/Impact: The proposed intervention has the potential to reduce ASCVD events in this population by more than a quarter and meet VA strategic priorities of: 1) improve timeliness of services; 2) focus resources more efficiently as well as address health systems research (HSR) research priorities: 1) patient centered care, care management, and health promotion; 2) healthcare access; 3) aging; 4) virtual care.

Innovation: The study is innovative: Cascade Model. By leveraging the HIV treatment cascade model, the investigators will create a pathway for ASCVD risk reduction to be added into widespread quality improvement initiatives. Stakeholder-engaged design process. The investigators will employ stakeholder-engaged research methods to ensure the intervention meets the needs of patients and healthcare providers. Multi-component nurse-led intervention. While each of the components of the intervention have an evidence base, they have not been tested together in an HIV context. Telehealth. The investigators will use VA Video Connect (VVC) to monitor CVD risk factors.

Specific Aims: Aim 1a: Conduct qualitative interviews with Veterans and healthcare providers to ascertain perceptions regarding HIV and CVD risk reductions to inform intervention adaptation.

Aim 1b: Adapt the intervention to the VA HIV clinic context with key stakeholder input.

Aim 2: Evaluate the 12-month efficacy of a nurse intervention to improve systolic blood pressure in Veterans with HIV. Hypothesis: The investigators hypothesize that the intervention will result in a clinically significant 6mmHg reduction in SBP over 12 months compared to those receiving [enhanced education + usual care] only. Aim 3: Conduct an evaluation of the prevention nurse intervention. Exploratory aim: If effective, [the investigators will conduct a budget impact analysis] and simulate 10-year cost-effectiveness of the nurse intervention.

Methodology: The investigators will conduct qualitative interviews with care team and Veterans to adapt the intervention in an iterative design process. The investigators will then conduct a RCT to evaluate an intervention to reduce ASCVD risk. The study will be conducted in 3 clinics among HIV+ Veterans (n=300) on suppressive antiretroviral therapy (ART) with confirmed SBP >140 mmHg, stratified by clinic site and randomized 1:1 to intervention vs. education control. The intervention will involve 4 evidence-based components based on the investigators' prior studies and adapted to Veterans with HIV: (1) nurse-led care coordination, (2) nurse-managed medication and adherence support (3) home BP monitoring, and (4) administered VA Video Connect (VVC). The education control will receive enhanced education and usual care. Primary outcome: difference in 12-month systolic BP in the intervention arm vs control. Secondary outcome: 12-month difference in non-HDL cholesterol. The investigators will use a mixed-methods design to evaluate fidelity, dose delivered/received, reach, recruitment, and context of the intervention.

Implementation/Next Steps: The investigators designed the intervention with downstream implementation in view. This includes: a fully remote delivery of the intervention to facilitate access and widespread implementation, and guidance for selection of nurses with education / experience levels that match those of health coaches delivering interventions within the VA. The investigators will work with operational partners from the Office of Connected Care and Office of HIV/AIDS care regarding implementation plans. The investigators will disseminate a clinical program, including scripts, and description of all intervention processes, to facilitate implementation within the VA.

ELIGIBILITY:
Inclusion Criteria:

1. Age => 18 years
2. Confirmed HIV+ diagnosis
3. Undetectable HIV viral load: defined as the most recent HIV viral load < 200 copies/mL, checked within the past 18 months (assessed via chart abstraction)
4. Hypertension: defined as the average of 4 most recent outpatient BP measurements in the last 18 months to show systolic BP 130 and/or diastolic 90 mmHg (assessed via chart abstraction)
5. Veteran at one of the sites participating in the study
6. Regular access to a computer, tablet or smart phone device with internet.

Exclusion Criteria:

1. Severely hearing or speech impaired, or other disability that would limit participation
2. In a nursing home at baseline and/or any long-term care facility. Individuals will be censored at the point of entering nursing home care
3. In-patient psychiatric care
4. Diagnosis of dementia or active psychosis
5. Terminal illness with life expectancy < 4 months (ex. Metastatic cancer, Hospice care)
6. Recent (<90day) hospitalization for coronary artery bypass surgery (CABG), myocardial infarction (MI), stroke)
7. Pregnant, breast-feeding, or planning a pregnancy during the study period
8. Planning to move out of the area in the next 12 months.
9. No reliable access to telephone services

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 305 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2025-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hayden B Bosworth, PhD, Principal Investigator — Durham VA Medical Center, Durham, NC; Puja Van Epps, MD, Principal Investigator — Louis Stokes VA Medical Center, Cleveland, OH
Locations (4):
- United States (4):
  - Atlanta VA Medical and Rehab Center, Decatur, GA, Decatur, Georgia
  - Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD, Baltimore, Maryland
  - Durham VA Medical Center, Durham, NC, Durham, North Carolina
  - Louis Stokes VA Medical Center, Cleveland, OH, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: Yes
Publications from this research will be made available to the public through the National Library of Medicine PubMed Central website within one year after the date of publication and study results will be available on Clinical Trials.gov within 1 year of the final follow-up with last study participant. A local privacy officer and study statistician will certify that the dataset contains no protected health information (PHI) prior to distribution. Data will be provided to requester in electronic form. Final data sets will be maintained locally until enterprise-level resources become available for long-term storage and access.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available within 1 year of the final follow-up with the last study participant.
Access Criteria: Guidance on request and distribution processes will be provided by the VA Office of Research and Development (ORD).

REFERENCES:
- [Result] Schexnayder J, Perry KR, Sheahan K, Majette Elliott N, Subramaniam S, Strawbridge E, Webel AR, Bosworth HB, Gierisch JM. Team-Based Qualitative Rapid Analysis: Approach and Considerations for Conducting Developmental Formative Evaluation for Intervention Design. Qual Health Res. 2023 Jul;33(8-9):778-789. doi: 10.1177/10497323231167348. Epub 2023 Jun 6. PMID 37278662
- [Result] Musoke L, Bosworth HB, Dickson C, Gentry P, Strawbridge E, Subramaniam S, Gierisch J, Smith V, Woolson S, Pura J, Amutuhaire W, Naggie S, Schexnayder J, Hall K, Longenecker CT, Harris NM, Rogers C, Van Epps P; for V-EXTRA-CVD Group. A telehealth-delivered intervention to extend the veteran HIV treatment cascade for cardiovascular disease prevention: V-EXTRA-CVD study protocol for a randomized controlled trial. HIV Res Clin Pract. 2023 Dec;24(1):2261747. Epub 2023 Oct 6. PMID 37800987

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: While 305 participants were consented and randomized to an arm, 4 withdrew and did not complete the baseline assessment.
  301 is the number that completed baseline assessment and will therefore be used as the baseline analytic population for the study.
Period: Overall Study
Arm/Group | Intervention Group | Education Control Group
Started | 152 | 149
Completed | 119 | 123
Not Completed | 33 | 26
Not completed — Withdrawal by Subject | 12 | 4
Not completed — Lost to Follow-up | 17 | 18
Not completed — 12month BP not collected | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Education Control Group | Total
Number analyzed (Participants) | 152 | 149 | 301
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.1 (9.6) | 61.4 (9.4) | 61.8 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 11 | 23
  Male | 140 | 138 | 278
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 10 | 18
  Not Hispanic or Latino | 139 | 136 | 275
  Unknown or Not Reported | 5 | 3 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 118 | 115 | 233
  White | 17 | 21 | 38
  More than one race | 9 | 11 | 20
  Unknown or Not Reported | 5 | 2 | 7
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 152 | 149 | 301
Education [Count of Participants; unit: Participants]
  High school or less | 39 | 41 | 80
  Some college or trade school | 69 | 62 | 131
  College graduate or higher | 44 | 46 | 90
Employment [Count of Participants; unit: Participants]
  Employed | 61 | 58 | 119
  Unemployed | 35 | 38 | 73
  Retired | 56 | 53 | 109

OUTCOME MEASURES:

1. Primary Outcome: Mean Systolic Blood Pressure
Description: Mean BP is calculated as the average of 3 BP measurements. Collected during BP outcome assessment conducted at interviews.
Time Frame: Baseline
Population: The randomized participants who completed the baseline assessment
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Intervention Group | Education Control Group
Number analyzed (Participants) | 152 | 149
mmHg | 134.6 (17.3) | 133.3 (15.5)

2. Primary Outcome: Mean Systolic Blood Pressure
Description: as for outcome 1
Time Frame: 4 months
Population: Enrolled participants who attended the in-person 4 month outcome assessment visit and had BP taken by study personnel.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Intervention Group | Education Control Group
Number analyzed (Participants) | 123 | 115
mmHg | 129.7 (14.6) | 129.6 (14.3)

3. Primary Outcome: Mean Systolic Blood Pressure
Description: as for outcome 1
Time Frame: 8 months
Population: Enrolled participants who attended the in-person 8 month outcome assessment visit and had BP taken by study personnel.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Intervention Group | Education Control Group
Number analyzed (Participants) | 107 | 109
mmHg | 130.4 (14.7) | 130.5 (16.6)

4. Primary Outcome: Mean Systolic Blood Pressure
Description: as for outcome 1
Time Frame: 12 months
Population: Enrolled participants who attended the in-person 12 month outcome assessment visit and had BP taken by study personnel.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Intervention Group | Education Control Group
Number analyzed (Participants) | 119 | 123
mmHg | 130.5 (13.4) | 130.6 (17.5)

5. Secondary Outcome: Non-HDL Cholesterol
Description: Non-HDL Cholesterol will be calculated by "Total Cholesterol - HDL Cholesterol" and will be collected by lab personnel during outcome assessments. It is measured in milligrams per deciliter (mg/dL)
Time Frame: Baseline
Population: The number of enrolled participants who visited the lab during their outcome assessment period and had blood lipids measured.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Intervention Group | Education Control Group
Number analyzed (Participants) | 151 | 148
mg/dL | 118.0 (42.6) | 120.9 (38.3)

6. Secondary Outcome: Non-HDL Cholesterol
Description: as for outcome 5
Time Frame: 4 months
Population: The number of enrolled participants who visited the lab during their 4 month outcome assessment period and had blood lipids drawn.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Intervention Group | Education Control Group
Number analyzed (Participants) | 125 | 120
mg/dL | 114.1 (51.0) | 115.4 (34.8)

7. Secondary Outcome: Non-HDL Cholesterol
Description: as for outcome 5
Time Frame: 8 months
Population: The number of enrolled participants who visited the lab during their 8 month outcome assessment period and had blood lipids drawn.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Intervention Group | Education Control Group
Number analyzed (Participants) | 108 | 113
mg/dL | 111.7 (42.9) | 116.4 (37.0)

8. Secondary Outcome: Non-HDL Cholesterol
Description: as for outcome 5
Time Frame: 12 months
Population: The number of enrolled participants who visited the lab during their 12 month outcome assessment period and had blood lipids drawn.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Intervention Group | Education Control Group
Number analyzed (Participants) | 123 | 127
mg/dL | 110.8 (39.7) | 115.2 (38.6)

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Intervention Group | Education Control Group
All-Cause Mortality (participants affected / at risk) | 3/152 | 1/149
Serious Adverse Events (participants affected / at risk) | 18/152 | 16/149
Other Adverse Events (participants affected / at risk) | 0/152 | 0/149
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention Group (N=152) | Education Control Group (N=149)
Gastroenteritis (Gastrointestinal disorders) | 0 | 2 (2)
Acute knee pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Chest pain hospitalization (Cardiac disorders) | 2 (2) | 2 (2)
Congestive Heart Failure Exacerbation (Cardiac disorders) | 3 (8) | 0 (0)
COVID hospitalization (Infections and infestations) | 1 (2) | 0 (0)
Defibrillator placement (Cardiac disorders) | 0 (0) | 1 (1)
Elective surgery (Surgical and medical procedures) | 2 (2) | 2 (2)
Falls (General disorders) | 1 (2) | 0 (0)
Gallbladder-related hospitalization (Hepatobiliary disorders) | 0 (0) | 1 (1)
Gastroenteritis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Inpatient rehab (Social circumstances) | 0 (0) | 1 (1)
Iron deficiency anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lithotripsy (Surgical and medical procedures) | 1 (1) | 0 (0)
Liver biopsy (Hepatobiliary disorders) | 0 (0) | 1 (1)
Orthostasis (General disorders) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)
Prostatectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Psychiatric admission (Psychiatric disorders) | 0 (0) | 1 (1)
Renal failure/injury (Renal and urinary disorders) | 2 (2) | 1 (1)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
UTI (Renal and urinary disorders) | 0 (0) | 1 (1)
Stent placement (Cardiac disorders) | 1 (1) | 0 (0)
Death (General disorders) | 3 (3) | 1 (1)

LIMITATIONS AND CAVEATS:
Recruitment challenges led to adjustments in inclusion criteria prior to study start, which affected baseline systolic blood pressure levels. The study was designed to evaluate systolic blood pressure (SBP) outcomes, not exploratory subgroup analyses.

The generalizability is limited to VA-based HIV populations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2024-09-09): https://cdn.clinicaltrials.gov/large-docs/89/NCT04545489/Prot_001.pdf
  • Statistical Analysis Plan (2025-06-06): https://cdn.clinicaltrials.gov/large-docs/89/NCT04545489/SAP_002.pdf
  • Informed Consent Form (2022-06-09): https://cdn.clinicaltrials.gov/large-docs/89/NCT04545489/ICF_000.pdf